CLINICAL TRIAL: NCT04808375
Title: Risk Factors for Pregnancy-induced Hypertension in Pregnant Patients Undergoing Cesarean Section: a Retrospective Study
Brief Title: Risk Factors for Pregnancy-induced Hypertension in Pregnant Patients Undergoing Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20210303
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Adverse Maternal and Neonatal Outcomes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
After Institutional Review Board approval, we performed a retrospective cohort study among all women presenting for pregnancy-induced hypertension under Cesarean section in Renji Hospital Affiliated to Shanghai Jiaotong University from January 2013 to January 2020.Perioperative data were collected, including preoperative general condition, laboratory examination, auxiliary examination (blood routine, blood coagulation, liver and kidney function, electrocardiogram, cardiac ultrasound, etc.), perioperative indicators, postoperative laboratory examination (blood routine, blood coagulation, liver and kidney function, etc.), postoperative follow-up and satisfaction survey of patients.

ELIGIBILITY:
Inclusion Criteria:

* all women presenting for pregnancy-induced hypertension in Renji Hospital Affiliated to Shanghai Jiaotong University from January 2013 to January 2020 cesarean section operation

Exclusion Criteria:

* no

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all women presenting for pregnancy-induced hypertension in Renji Hospital Affiliated to Shanghai Jiaotong University from January 2013 to January 2020 cesarean section operation
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-03-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Adverse maternal outcomes | 42 days after delivery
  Adverse maternal outcomes were evaluated individually and as a composite and included number of acute kidney injury (serum creatinine >1.1 mg/dL or oliguria), number of blood transfusion, number of eclampsia, rate of intensive care unit (ICU) admission, number of postpartum hemorrhage, or pulmonary edema.(From date of randomization until the date of discharged from hospital, whichever came first, assessed up to 40 weeks").
Adverse neonatal outcomes | 42 days after delivery
  Number of neonatal outcomes included preterm birth (PTB; <37 weeks), Number of neonatal ICU (NICU) admission, number of neonatal intubation, and number of respiratory distress syndrome.（From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40weeks）.(From the date of birth until the date of discharged from hospital, whichever came first, assessed up to 5 weeks").

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China